CLINICAL TRIAL: NCT00059501
Title: Cortical Control of Postural Stability in the Elderly
Brief Title: Postural Control in the Elderly
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030165; 03-N-0165
Record Dates: First submitted 2003-04-26; First posted 2003-04-28 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Musculoskeletal Physiology; Healthy
Keywords: Postural Stability; EEG; Aging; Falls; Healthy Volunteer; HV

SUMMARY:
This study will examine loss of balance in the elderly. Falls due to balance problems are a major health issue in older people, often resulting in bone fractures and other bodily injuries, and functional decline. In addition, the fear of falling leads some elderly people to restrict their movements and social activities, causing depressed moods and decreased enjoyment of life. Risk factors for falling in the elderly include some standing positions in which older people usually experience balance problems, such as leaning forward or backward. This study will examine these unstable positions and the brain mechanisms associated with loss of balance in the elderly.

Normal volunteers between 20 and 90 years of age may be eligible for this study. Candidates must be in good health, with no difficulties in performing activities of daily living, and must be able to walk for at least 400 meters (1/4 mile). They will be screened with a medical history, physical examination, and blood tests.

Participants will undergo the following three experiments:

* Movement task: The subject stands on a platform with markers placed at different parts of the body to record body movements. A cap with electrodes (metal disks) is placed on the head for electrocardiographic (EEG) recording of the electrical activity of the brain (brain waves) during the experiment. The positions of the feet on the platform are measured. While standing on the platform, the subject leans forward and backward as far as possible without losing balance. (Subjects are secured in a safety harness to prevent actual falls.) The task is repeated 5 times. The experiment lasts up to 2 hours.
* Postural response task: This study is identical to the first, except that the subject does not voluntarily lean forward and backward, but is pushed with a device to cause forward and backward movements. The experiment lasts 1 to 2 hours.
* Perceptual task: The subject sits in front of a computer screen and watches the postural movements of a human body model in forward and backward directions. When the subject recognizes an unstable position in the movements, he or she presses a computer mouse. An EEG records brain activity during the task, which lasts up to 2 hours.

DETAILED DESCRIPTION:
A number of studies have explored the role of visual, vestibular and somatosensory systems in the control of upright posture. However, the cortical control of postural stability, in general, and the role of higher cognitive function in assessment of postural stability, in specific, has been less studied. It is well established that certain features of postural control change during the advancing years of life so that the stability of posture can be a problem in the elderly. However, neural mechanisms of postural stability that decline with age and make older adults more prone to falling have not been identified specifically. To characterize specific causes of falling in the elderly in problematic, because human posture is a product of an extremely complex dynamical system and like any other physical activity undergoes dramatic changes in organization throughout the life-span. In our previous research we showed the existence of specialized neural detectors that are embodied in spatiotemporal patterns of brain activiation (Slobounov et al., 200) capable of discrimination the unstable postures in dynamic situations. We propose that these neural detectors may deteriorate with aging, which result in difficulty to (a) initiate compensatory postural adjustments when balance is in danger, and (b) to discriminate relevant from irrelevant information in control of upright posture. This can be documented via changes in behavioral correlates of postural control and spatiotemporal patterns of the brain activation as a function of advanced age. Accordingly, the purpose of this study is to investigate the age-related cortical control of postural stability combining electroencephalography and postural control measures. This will be done when a subject physically approaches the postural stability boundary and when a subject solves a cognitive task identifying unstable postures in dynamic situations.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects will be enrolled in this balance study if they are within the range of 20-90 years old;

in good health;

report no difficulties or need for help in performing self-care or instrumental activities of daily living;

and are able to walk for at least 400 meters.

EXCLUSION CRITERIA:

We will be unable to study people who have substantial congitive impairment based on mental status screening tests;

history of cardiovascular disease (including angina, myocardial infarction, congestive heart failure, cerebro-vascular disease);

cancer;

neurological diseases;

birth defects;

kidney or liver disease;

gastrointestinal (G.I.) disease;

musculo-skeletal disorder (if they cause pathological weakness and/or chronic pain);

important sensory deficits and any conditions that precludes them from being tested with standard neurophyschological tests.

Pregnant women will be excluded from this study.

In addition, the following criteria are considered as markers of pathological conditions and are used as exclusion criteria for study enrollment:

1. HIV virus infection;
2. WBC greater than 12,000 ML;
3. Platelets less than 100,000 or greater than 600,000/ML;
4. Hemoglobin less than 11 gr/dl unless higher level can be ascribed to Gilbert's disease;
5. Abnormal level of SGOT and SGPT and alkaline phosphetase twice the norm serum concentration;
6. Corrected calcium less than 8.5 or 10.7 mg/dl;
7. Albumin less than 3.4 g/dl;
8. Shortness of breath while performing normal activities of daily living, such as walking or climbing stairs;
9. evidence or history of cancer;
10. absolute need for long term treatment with antibiotics, corticosteroids, immunosuppressors, H2 blockers and pain medications;
11. any severe psychiatric condition such as subjects with Axis I psychiatric diagnosis;
12. any condition that may preclude informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 2003-04; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Arfken CL, Lach HW, Birge SJ, Miller JP. The prevalence and correlates of fear of falling in elderly persons living in the community. Am J Public Health. 1994 Apr;84(4):565-70. doi: 10.2105/ajph.84.4.565. PMID 8154557
- [Background] Dunn JE, Rudberg MA, Furner SE, Cassel CK. Mortality, disability, and falls in older persons: the role of underlying disease and disability. Am J Public Health. 1992 Mar;82(3):395-400. doi: 10.2105/ajph.82.3.395. PMID 1531583
- [Background] Eeg-Olofsson O. Longitudinal developmental course of electrical activity of brain. Brain Dev. 1980;2(1):33-44. doi: 10.1016/s0387-7604(80)80006-4. PMID 7416440